CLINICAL TRIAL: NCT04716348
Title: Efficacy of Muscle Energy Technique on Forward Head Posture and Cervical Mobility in Visually Impaired Children
Brief Title: Muscle Energy Technique on Forward Head Posture and Cervical Mobility in Visually Impaired Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Egyptian Chinese University (Other)
Responsible Party: Principal Investigator, Noha Elserty, lecturer of physical therapy, Egyptian Chinese University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Egyptian Chinese University
Record Dates: First submitted 2021-01-11; First posted 2021-01-20 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Children With Visual Disabilities

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): suboccipital muscle energy technique
  Interventions: Procedure: muscle energy technique
- group B (Sham Comparator): sham muscle energy technique
  Interventions: Procedure: muscle energy technique

INTERVENTIONS:
Procedure: muscle energy technique — muscle energy technique for suboccipital muscles

SUMMARY:
Forward head posture is one of the most common postural deviation seen among visually impaired children and, it is characterized by hyperextension of upper cervical and flexion of lower cervical spine. These changes lead to muscle imbalance and resulting in weakness of the deep cervical flexors, shortening of the opposing cervical extensors and reduction in cervical range of motion. Muscle energy technique is a manual therapy technique using in the treatment of shortened muscles, muscle weakness, restricted joints range of motion. so this study aimed to investigate the efficacy of muscle energy technique on forward head posture and cervical mobility in visually impaired children.

DETAILED DESCRIPTION:
subjects will be allocated according to the inclusion and exclusion criteria from different schools for visually impaired children. They will be divided randomly into study group and control group. Study group will be participated in suboccipital muscle energy technique. Control group will be participated in sham technique. The duration of treatment for both groups will be 3 times/week for 6 weeks. Autodesk AutoCAD software will be used to analyze the measured angles and CROM will be used to assess cervical mobility

ELIGIBILITY:
Inclusion Criteria:

* Visual acuity will be 6/24, 6/36 and 6/60 after correction.
* Wearing glasses more than one year.
* Craniovertebral angle < 50°.
* Functional hearing.

Exclusion Criteria:

* Injury of cervical region (e.g: atlantoaxial instability).
* Cervical spine deformities or/disorders.
* History of previous cervical spine surgery.
* Rheumatic and congenital heart disease.
* Regular participation in any sport activities.
* Intellectual or/mental disabilities

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
change in craniovertebral angle | baseline pre intervention and immediately after the intervention
  analysis of craniovertebral angle form lateral view performed by AUTOCAD program
change of cervical range of motion | baseline pre intervention and immediately after the intervention
  measurement of cervical range of motion including cervical flexion, cervical extension, cervical side bending, and cervical rotation. these measurement will be applied by CROM device

CONTACTS AND LOCATIONS:
Overall Officials: Noha S Elserty, PhD, Principal Investigator — Lecturer of physical therapy- Egyptian Chinese University
Locations (1):
- Noha Elserty, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
supporting information that will be shared after publication of the study
Supporting Information: Study Protocol, SAP
Time Frame: after publishing the study